CLINICAL TRIAL: NCT02062645
Title: A Single-Arm Open-Label Multicenter Phase IV Clinical Trial to Explore the Blood Pressure Lowering Effect of Exforge® (Amlodipine/Valsartan: AMLO/VAL) in Hypertensive Patients
Brief Title: Study of Efficacy and Safety of CVAA489 in Hypertensive Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CVAA489ATR04
Record Dates: First submitted 2014-02-12; First posted 2014-02-14 (Estimated); Results first posted 2017-03-28 (Actual); Last update posted 2017-03-28 (Actual); Status verified 2017-02

CONDITIONS: Essential Hypertension
Keywords: essential hypertension
MeSH Terms: conditions — Essential Hypertension | interventions — Amlodipine, Valsartan Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- amlodipine/valsartan (Experimental): All patients will receive amlodipine/valsartan 5/160 mg daily in screening and up titrated to amlodipine/valsartan 10/160 mg daily at visit 2 (day 30) if their hypertension can not be controlled. The duration of treatment period is 8 weeks.
  Interventions: Drug: amlodipine/valsartan

INTERVENTIONS:
Drug: amlodipine/valsartan — Fixed combination of amlodipine and valsartan in tablet; 5/160/mg, 10/160 mg

SUMMARY:
The population that will be included in this study, will be regular Turkish hypertensive patients who are expected to consume sodium in high amounts. It is hypothesized that, in that population, amlodipine/valsartan will be effective at the same rate of blood pressure (BP) control rate as expected from literature.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, above 18 years of age
* Diagnosis of essential hypertension
* Newly diagnosed,
* Previously untreated, or Currently untreated (not on regular antihypertensive treatment during the previous at least 1-month period)
* Written informed consent

Exclusion Criteria:

* Known or suspected secondary hypertension
* eGFR lower than 30 mL/min
* Use of any other hypertension treatments during the enrollment and need for using the related treatments during the study phase
* History of hypersensitivity to any of the study drugs or to drugs of similar chemical classes. (i.e. valsartan, amlodipine, hydrochlorothiazide)
* History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.
* Use of other investigational drugs within 5 half-lives of enrollment, or within 30 days until the expected PD effect has returned to baseline, whichever is longer.Pregnant or nursing (lactating) women
* Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 115 (Actual)
Dates: Start 2014-02; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (8):
- Turkey (Türkiye) (8):
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Çanakkale
  - Novartis Investigative Site, Fatih / Istanbul
  - Novartis Investigative Site, Kinikli / Denizli
  - Novartis Investigative Site, Kocaeli
  - Novartis Investigative Site, Malatya
  - Novartis Investigative Site, Mersin
  - Novartis Investigative Site, Talas / Kayseri

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One hundred thirty patients were screened and 115 were enrolled into the trial.
Groups:
- Amlodipine/Valsartan: All patients received amlodipine/valsartan 5/160 mg daily at Day 0 and were up titrated to amlodipine/valsartan 10/160 mg daily at visit 2 (week 4) if their hypertension was not controlled. The duration of treatment period was 8 weeks.
Period: Overall Study
Arm/Group | Amlodipine/Valsartan
Started | 115
Completed | 100
Not Completed | 15
Not completed — Adverse Event | 2
Not completed — Protocol Violation | 8
Not completed — Lost to Follow-up | 5

BASELINE CHARACTERISTICS:
Population: The baseline population was the ITT (intent to treat) population defined as: met all entry criteria, received study drug and had at least one blood pressure measurement after Visit 1 (Day 0)
Arm/Group | Amlodipine/Valsartan
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.06 (11.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55
  Male | 45
Systolic blood pressure [Mean (Standard Deviation); unit: mmHG] | 164.3 (13.2)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 96.7 (12.7)
Heart rate [Mean (Standard Deviation); unit: beats/min] | 80.15 (10.00)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 31.19 (5.32)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Blood Pressure (BP) <140/90 mmHg at Week 4 and 8
Description: Control rate of BP defined as BP lower than 140/90 mmHg at office visits
Time Frame: At week 4 and 8
Population: The ITT (intent to treat) population defined as: met all entry criteria, received study drug and had at least one blood pressure measurement after Visit 1 (Day 0). One hundred patients had BP measurements at Visit 2 and 91 patients at Visit 3. LOCF (Visit 2 to Visit 3). Analysis performed both with original and imputed values
Measure: Number; unit: Percentage of Participants
Arm/Group | Amlodipine/Valsartan
Number analyzed (Participants) | 100
Percentage of Participants
  Week 4 Systolic (n=100) | 47.0
  Week 4 Diastolic (n=100) | 78.0
  Week 4 Overall Blood Pressure(n=100) | 45.0
  Week 8 Systolic(n=91) | 70.3
  Week 8 Diastolic (n=91) | 82.4
  Week 8 Overall Blood Pressure (n=91) | 67.0
  Week 8 Systolic (LOCF) (n=100) | 68.0
  Week 8 Diastolic (LOCF) (n=100) | 81.0
  Week 8 Overall Blood Pressure (LOCF) (n=100) | 65.0

2. Secondary Outcome: Systolic Blood Pressure (SBP) at Baseline, Week 4 and 8
Description: Change in systolic blood pressure measured in office from baseline at week 4 and 8.
Time Frame: baseline, week 4, week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Amlodipine/Valsartan
Number analyzed (Participants) | 100
mmHg
  Systolic blood pressure (SBP) Day 0 (n=100) | 164.3 (13.2)
  Systolic blood pressure (SBP) Week 4 (n=100) | 140.17 (14.05)
  Systolic blood pressure (SBP) Week 8 (n=91) | 134.04 (13.51)
  Systolic blood pressure (SBP) Week 8 LOCF (n=100) | 134.71 (13.37)
  Decrease in Systolic Week 4 (n=100) | 24.15 (18.18)
  Decrease in Systolic Week 8 (n=91) | 30.22 (18.25)
  Decrease in Systolic BP Week 8 LOCF (n=100) | 29.61 (17.81)

3. Secondary Outcome: Diastolic Blood Pressure (DBP) at Baseline, Week 4 and 8
Description: Change in diastolic blood pressure measured in office from baseline at week 4 and week 8.
Time Frame: baseline, week 4, week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Amlodipine/Valsartan
Number analyzed (Participants) | 100
mmHg
  Diastolic blood pressure (DBP) Day 0 (n=100) | 96.66 (12.68)
  Diastolic blood pressure (DBP) Week 4 (n=100) | 82.0 (9.88)
  Diastolic blood pressure (DBP) Week 8 (n=91) | 81.04 (8.66)
  Diastolic blood pressure (DBP) Week 8 LOCF (n=100) | 81.37 (8.69)
  Decrease in Diastolic BP Week 4 (n=100) | 14.66 (12.58)
  Decrease in Diastolic BP Week 8 (n=91) | 15.54 (13.19)
  Decrease in Diastolic BP Week 8 LOCF (n=100) | 15.29 (12.73)

4. Secondary Outcome: Percentage of Participants With High Sodium Intake and Blood Pressure (BP) <140/90 mmHg at Week 4 and 8
Description: Control rate of BP is defined as blood pressure lower than 140/90 mmHg at office visits in patients with high sodium intake (>100 mEq/day)
Time Frame: At week 4 and 8
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Amlodipine/Valsartan
Number analyzed (Participants) | 70
Percentage of participants
  Week 4 (n=70) | 68.6
  Week 8 (n=64) | 64.1
  Week 8 LOCF (n=70) | 62.9

5. Secondary Outcome: SBP and DBP in Patients With High Sodium Intake at Week 4 and 8
Description: Change in systolic and diastolic blood pressure measured in office from baseline at week 4 and 8.
Time Frame: At week 4 and 8
Population: All patients received amlodipine/valsartan 160/5 mg daily at Day 0 and were up titrated to amlodipine/valsartan 160/10 mg daily at visit 2 (week 4) if their hypertension can not be controlled. The duration of treatment period was 8 weeks.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Amlodipine/Valsartan
Number analyzed (Participants) | 70
mmHg
  SBP at Week 4 (n=70) | 140.01 (13.67)
  SBP at Week 8 (n=64) | 134.20 (13.24)
  SBP at Week 8 LOCF (n=70) | 134.84 (13.17)
  DBP at Week 4 (n=70) | 81.73 (10.26)
  DBP at Week 8 (n=64) | 81.23 (8.80)
  DBP at Week 8 LOCF (n=70) | 81.47 (8.91)

ADVERSE EVENTS:
Description: The safety population included data from patients who attended Visit 2 which was 110 patients.
Groups:
- Amlodipine/Valsartan: amlodipine/valsartan
Arm/Group | Amlodipine/Valsartan
Serious Adverse Events (participants affected / at risk) | 3/110
Other Adverse Events (participants affected / at risk) | 76/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Amlodipine/Valsartan (N=110)
Death (General disorders) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Amlodipine/Valsartan (N=110)
Anaemia (Blood and lymphatic system disorders) | 7
Aortic valve incompetence (Cardiac disorders) | 10
Diastolic dysfunction (Cardiac disorders) | 5
Left atrial dilatation (Cardiac disorders) | 4
Left ventricular dysfunction (Cardiac disorders) | 34
Left ventricular hypertrophy (Cardiac disorders) | 30
Mitral valve incompetence (Cardiac disorders) | 16
Tricuspid valve incompetence (Cardiac disorders) | 8
Nausea (Gastrointestinal disorders) | 3
Oedema peripheral (General disorders) | 3
Blood uric acid increased (Investigations) | 3
Electrocardiogram abnormal (Investigations) | 3
Urine sodium increased (Investigations) | 8
Microalbuminuria (Renal and urinary disorders) | 6
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 3
Aortic aneurysm (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial